CLINICAL TRIAL: NCT06659692
Title: Pharmacokinetics of Follicle-stimulating Hormone and Human Chorionic Gonadotrophin Following Multiple Daily Subcutaneous Injections of Gonadotropins-IBSA in Pituitary Down-regulated Female Subjects.
Brief Title: Pharmacokinetics of FSH and hCG Following Multiple Dose of Gonadotropins-IBSA.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23CDN-FCG09
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Stimulation; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gonadotropins 150 IU (Experimental): 150 IU daily for 7 days.
  Interventions: Drug: Gonadotropins Subcutaneous
- Gonadotropins 300 IU (Experimental): 300 IU daily for 7 days
  Interventions: Drug: Gonadotropins Subcutaneous

INTERVENTIONS:
Drug: Gonadotropins Subcutaneous — Gonadotropins s.c. multiple dose

SUMMARY:
Pharmacokinetics of FSH and hCG after multiple subcutaneous injection of Gonadotropins-IBSA.

ELIGIBILITY:
Inclusion Criteria:

1. Female of childbearing potential, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤45 years of age, with BMI >18.5 and <32.0 kg/m2 and body weight ≥45.0 kg.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Use of a COC containing at least 20 µg of ethinyl estradiol for at least 3 months prior to screening and willing to keep using the same oral contraceptive until the end of the study. The usual regimen (with hormone-free interval or continuous dosing) will be allowed until Day -1. Subjects must agree to take the COC in a continuous manner (no hormone-free interval) from Day 1 to Day 36.
4. Females who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized for at least 3 months prior to dosing) must be willing to use a male condom with intravaginally applied spermicide or total abstinence from heterosexual intercourse (when this is in line with the preferred and usual lifestyle of the subject) from screening and throughout the study and for 30 days after the last study drug administration.
5. Able to understand the study procedures and provide signed informed consent to participate in the study

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening.
2. Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.
3. Positive pregnancy test or lactating subject.
4. Positive urine drug screen, urine cotinine test, or alcohol breath test.
5. Known allergic reactions to FSH, hCG, other gonadotropins, or other related drugs, or to any excipient in the formulation.
6. Clinically significant ECG abnormalities or vital signs abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
7. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
8. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
9. FSH levels > 4 IU/L at admission in each period.
10. Presence of ovarian cysts > 10 mm in size or clinically significant ovarian enlargement at admission (Day 19).
11. Clinically significant history of an abnormal menstrual cycle.
12. Abnormal Pap smear prior to administration of the study drug (result is valid for 12 months).
13. History of ovarian cysts or enlargement.
14. History or presence of polycystic ovary syndrome.
15. Presence of undiagnosed vaginal and/or urinary tract bleeding.
16. History or presence of sex hormone dependent tumours of reproductive tract and accessory organs.
17. History of hypothalamus or pituitary gland tumours.
18. Personal history or strong family history (first degree relative) of coagulation disorders such as thromboembolic diseases (e.g., thrombophlebitis, pulmonary embolism or coagulation factors deficiency).
19. History of rare hereditary galactose and/or lactose intolerance (e.g., congenital lactase deficiency [CLD] or glucose-galactose malabsorption [GGM]).
20. Tattoos covering the potential study drug injection site or any skin conditions that would prevent the injection (e.g., psoriasis, major scar, etc.).
21. Use of medications for the timeframes specified below, except for the subject's prescribed COC and medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. depot injection or implant of any drug within 3 months prior to study drug administration;
    2. prescription medications within 14 days prior to study drug administration;
    3. any vaccines, including COVID-19 vaccine, within 14 days prior to study drug administration;
    4. over-the-counter (OTC) products and natural health products (including herbal remedies such as St. John's wort, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to study drug administration, with the exception of the occasional use of acetaminophen (up to 2 g daily);
22. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
23. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
24. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Primary PK endpoints | until 240 hours post dose.
  Day 20: AUC0-24
Primary PK endpoints | until 240 hours post dose.
  Day 20:Cmax: to assess the bioavailability of the test product in terms of rate (baseline-corrected, dose-normalised Cmax) of Gonadotropins-IBSA absorption after multiple s.c. injection to healthy female subjects.
Primary PK endpoints | until 240 hours post dose.
  Day 20: Tmax (Time to achieve Cmax)
Primary PK endpoints | until 240 hours post dose.
  Day 26: AUC0-24
Primary PK endpoints | until 240 hours post dose.
  Day 26: Cmax: to assess the bioavailability of the test product in terms of rate (baseline-corrected, dose-normalised Cmax) of Gonadotropins-IBSA absorption after multiple s.c. injection to healthy female subjects.
Primary PK endpoints | until 240 hours post dose.
  Day 26: Tmax (Time to achieve Cmax)
Primary PK endpoints | Through the duration of the study
  Accumulation potential: Rac

SECONDARY OUTCOMES:
Inhibin B | until 240 hour post last dose
  Analysis of Inhibin B
Estradiol (E2) | until 240 hour post last dose.
  Analysis of Estradiol (E2)
Number of Follicle | After seven days of treatment
  Follicle growth
Adverse events (AEs) | From the signature of the Informed Consent until the end of the study.
  Percentage of subjects with any AEs
Immunogenicity | At pre-dose on Day 20.
  Incidence of anti-FSH antibodies be analyzed only for subjects with ADA positive results.
Immunogenicity | 240 hours post-last dose
  Incidence of anti-FSH antibodies be analyzed only for subjects with ADA positive results.
Immunogenicity | 576 hours post last dose
  Incidence of anti-FSH antibodies
Immunogenicity | At pre-dose on Day 20
  Incidence anti-hCG antibodies
Immunogenicity | 240 hours post-last dose and 576 hours post last dose.
  Incidence anti-hCG antibodies
Immunogenicity | 576 hours post last dose.
  Incidence anti-hCG antibodies
Immunogenicity | Only for subjects with ADA positive
  Neutralizing antibodies (NAbs)

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No